CLINICAL TRIAL: NCT01435044
Title: QUANTUM: An International, Multi-center, Blinded, Randomized Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Administration of Regimens Containing PSI-352938, PSI-7977, and Ribavirin in Patients With Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Safety Study of Regimens of Sofosbuvir, GS-0938, and Ribavirin in Patients With Chronic Hepatitis C Infection
Acronym: QUANTUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P2938-0721
Record Dates: First submitted 2011-09-09; First posted 2011-09-15 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; Chronic; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — Sofosbuvir; PSI 352938; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- SOF+RBV 12 Weeks (Experimental): Participants were randomized to receive sofosbuvir plus RBV plus placebo to match GS-0938 for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV
- SOF+RBV 24 Weeks (Experimental): Participants were randomized to receive sofosbuvir plus RBV plus placebo to match GS-0938 for 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV
- GS-0938 Alone (Experimental): Participants were randomized to receive GS-0938 plus placebo to match sofosbuvir for up to 24 weeks.
  Interventions: Drug: GS-0938; Drug: Placebo to match sofosbuvir
- GS-0938+SOF (Experimental): Participants were randomized to receive GS-0938 plus sofosbuvir for up to 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: GS-0938
- GS-0938+SOF+RBV (Experimental): Participants were randomized to receive GS-0938 plus sofosbuvir plus RBV for up to 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: GS-0938; Drug: RBV
- Placebo (Experimental): Deferred start group: Participants were randomized to receive placebo to match GS-0938 plus placebo to match sofosbuvir for 24 Weeks.
  Interventions: Drug: Placebo to match sofosbuvir; Drug: Placebo to match GS-0938
- Retreatment Group - SOF+RBV 24 Weeks (Experimental): After discontinuing a regimen containing GS-0938, participants received sofosbuvir plus RBV for up to 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg (2 × 200 mg tablets) administered orally once daily
  Other Names: Sovaldi™; GS-7977; PSI-7977
  Arms: GS-0938+SOF; GS-0938+SOF+RBV; Retreatment Group - SOF+RBV 24 Weeks; SOF+RBV 12 Weeks; SOF+RBV 24 Weeks
Drug: GS-0938 — GS-0938 300 mg (3 × 100 mg tablets) administered orally once daily
  Other Names: PSI-352938
  Arms: GS-0938 Alone; GS-0938+SOF; GS-0938+SOF+RBV
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Ribasphere®
  Arms: GS-0938+SOF+RBV; Retreatment Group - SOF+RBV 24 Weeks; SOF+RBV 12 Weeks; SOF+RBV 24 Weeks
Drug: Placebo to match sofosbuvir — Placebo to match sofosbuvir administered orally once daily
  Arms: GS-0938 Alone; Placebo
Drug: Placebo to match GS-0938 — Placebo to match GS-0938 administered orally once daily
  Arms: Placebo

SUMMARY:
This study was designed to assess the safety and efficacy of multiple interferon-free treatment regimens of sofosbuvir (Sovaldi™; GS-7977; PSI-7977) and GS-0938 (PSI-352938) alone and in combination, with and without ribavirin (RBV). Each regimen was to be evaluated over 12 and 24 weeks to identify the optimal duration of therapy to maximize the benefit (sustained virologic response [SVR]) versus risk (safety and resistance).

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV-infection
* Naive to all HCV antiviral treatment
* Otherwise healthy patients

Exclusion Criteria:

* Positive test at Screening for HBsAg, anti-HBc IgM Ab, or anti-HIV Ab
* History of any other clinically significant chronic liver disease
* Medical history which the investigator considers the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with sustained virologic response (SVR) 12 weeks after discontinuation of study drug (SVR12) | Post-treatment Week 12
  SVR12 was defined as HCV RNA < LLOQ 12 weeks after the last dose of all study drugs.

SECONDARY OUTCOMES:
Percentage of Participants Who Experienced Adverse Events | Baseline to Week 24 plus 30 days
  Adverse events (AEs) were summarized across the participant population. A participant was counted once if they had a qualifying event.
Change from baseline in HCV RNA | Baseline to Week 12
Percentage of Participants With HCV RNA < LLOQ during treatment | Baseline to Week 12
Percentage of Participants With ALT Normalization | Baseline to post-treatment Week 4
  ALT normalization was defined as ALT > ULN at baseline and ALT ≤ ULN at a subsequent visit.
Percentage of participants with SVR at 4 and 24 weeks after discontinuation of study drug (SVR4; SVR24) | Post-treatment Weeks 4 and 24
  SVR4 and SVR24 was defined as HCV RNA < LLOQ 4 and 24 weeks after the last dose of all study drugs, respectively.
Percentage of Participants Who Developed Resistance to Sofosbuvir | Baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Hyland, DPhil, Study Director — Gilead Sciences
Locations (44):
- United States (42):
  - Alabama Liver & Digestive Specialists, Montgomery, Alabama
  - Bakersfield, California
  - Coronado, California
  - La Mesa, California
  - Los Angeles, California
  - CLI, Los Angeles, California
  - UCSD Antiviral Research Center, San Diego, California
  - eStudy Site, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Denver, Colorado
  - Engelwood, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Washington D.C., District of Columbia
  - Avail Clinical Research, DeLand, Florida
  - University of Florida Hepatology, Gainesville, Florida
  - University of Miami Center for Liver Diseases, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Advanced Research Institute, Trinity, Florida
  - South Florida Center of Gastroenterology, Wellington, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Digestive Health Services, Downers Grove, Illinois
  - Investigative Clinical Research, Annapolis, Maryland
  - Baltimore, Maryland
  - ID Care, Hillsborough, New Jersey
  - Concorde Medical Group, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Ashville Gastroenterology Associates, Ashville, North Carolina
  - Carolina's Center for Liver Disease, Statesville, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Gastro One, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Central Texas Clinical Research, Austin, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Puerto Rico (2):
  - San Juan, Puerto Rico
  - Fundacion de Investigacion de Diego, San Juan